CLINICAL TRIAL: NCT03342950
Title: The Effects of Topical Treatment With Clonidine + Pentoxifylline in Patients With Neuropathic Pain
Acronym: TTNP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment due to the COVID-19 pandemic
Sponsor: Terence J. Coderre (Other)
Collaborators: The Louise And Alan Edwards Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Terence J. Coderre, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A03-M45-15B
Record Dates: First submitted 2017-11-01; First posted 2017-11-17 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Neuralgia Peripheral
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug group (Active Comparator): Treatment with the topical solution of clonidine + pentoxifylline (0.1%/5%)
  Interventions: Drug: Topical Solution
- Placebo group (Placebo Comparator): Treatment with placebo solution with out active drug ingredients
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Topical Solution — Topical Solution of Clonidine (0.01%) + Pentoxifylline (5%) in anhydrous ethanol (6.5%), polyethylene glycol 400 (20%), propylene glycol (53.5%), and oleyl alcohol (20%)
  Arms: Active drug group
Drug: Placebos — Topical Solution of anhydrous ethanol (6.5%), polyethylene glycol 400 (20%), propylene glycol (53.5%), and oleyl alcohol (20%)
  Arms: Placebo group

SUMMARY:
Microvascular dysfunction underlies pain in different animal models of neuropathic pain. Pentoxifylline is a phosphodiesterase inhibitor that reduces cyclic adenosine monophosphate (cAMP) hydrolysis, enhances blood flow and reduces platelet aggregation, decreases blood viscosity, and increases the flexibility of red blood cells, all of which relieve microvascular dysfunction. Clonidine is an α2-adrenergic receptor agonist that decreases sympathetic outflow from the brainstem, vascular reactivity and has direct peripheral vasodilatory action. Topical combination of pentoxifylline and clonidine produced significant antiallodynic effects in rat models of neuropathic pain with sciatic nerve injury, painful diabetic neuropathy, and chemotherapy-induced painful neuropathy. In healthy volunteers with an experimentally-induced surrogate for neuropathic pain: post-capsaicin tourniquet exposure, the topical combination reduced areas of dynamic allodynia and mechanical hyperalgesia, in addition to reducing post-capsaicin ischemic pain.

This study will investigate if the same topical combination of clonidine + pentoxifylline will relieve pain in patients with neuropathic pain following traumatic injuries of peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, aged 18-70;
2. An average spontaneous pain level of at least 4 on an 11-point numerical rating pain score (0= no pain, 10= worst pain possible) on at least 3 days during the week prior to the study;
3. The existence of tactile allodynia, as a sign of chronic pain, following a traumatic peripheral nerve injury;
4. Ability to communicate in English or in French;
5. Willing and able to sign an informed consent;
6. Stable pain disease with no anticipated change in treatment in the next 5 weeks.
7. Female subjects of childbearing potential must agree to use effective method of contraception during the study period. Female subjects who utilize a hormonal contraceptive as one of their birth control methods must have consistently used the same method for at least three months prior to study drug dosing.

Exclusion Criteria:

1. Diabetes mellitus necessitating antihyperglycemic treatment or any other endocrine disease;
2. Any liver disease, resulting in aspartate aminotransferase (AST) levels greater than 3 times the normal values, or kidney disease, resulting in creatinine levels greater than 133 µmol/L;
3. Hypertension or taking of anti-hypertensive medication;
4. Malignant disease or taking of chemotherapeutic agents;
5. Known diagnosis of angina pectoris, arrhythmias, congestive heart failure or peripheral arterial disease;
6. Pregnancy or breast feeding. Female patients of child-bearing age must have a negative urine pregnancy test;
7. Known allergic reaction to clonidine or pentoxifylline;
8. Presence of major depression, bipolar affective disorder or schizophrenia;
9. Presence of a severe medical condition, or condition known to affect peripheral circulation (intermittent claudication, peripheral arterial disease, Raynaud's syndrome);
10. any medication that interacts with clonidine or pentoxifylline [e.g. cardiovascular drugs such as angiotensin converting enzyme (ACE) inhibitors, alpha blockers (prazosin, terazosin or doxazosin), beta blockers (atenolol, metoprolol, propranolol), neuroleptics (butyrophenones, phenothiazines, thioxanthenes), calcium channel blockers (verapamil, diltiazem) and non-cardiovascular drugs such as diuretics, thyroxine, monoamine oxidase inhibitors and selective serotonin reuptake inhibitors (SSRIs), as well as vitamin K antagonists/blood thinners, such as warfarin];
11. any medical condition that might be impacted by clonidine or pentoxifylline, such as cardiovascular disease, cardiac rhythm disorders (atrial-ventricular blockade or conduction abnormalities), orthostatic regulation disturbances, disorders of cerebral perfusion, chronic renal failure; sinus node dysfunction, or a recent cerebral and/or retinal haemorrhage.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale (VAS) score of spontaneous pain intensity | Scores recorded on pain diary on trial day 1, day 14 , day 21 and day 35 will be used
  This will be an evaluation of patients' daily spontaneous pain recorded on a pain diary. The visual analogue scale is a 100 millimetre line with the words "no pain" and "worst pain possible" on the left and right of it respectively. The patients will indicate their level of pain by marking on the line. The position of the mark on the line from the left end to the right will be measured in millimetres to obtain level of pain severity (The higher the VAS score the more severe the pain) . Change in VAS score will be obtained by comparing the difference between scores recorded on trial day 1 versus trial day 14 and trial day 21 versus trial day 35.
Change in visual analogue scale (VAS) score of dynamic mechanical allodynia (DMA) | Scores obtained from tests performed on trial day 1, day 14, day 21 and day 35 will be used.
  The degree of dynamic mechanical allodynia will be determined by stroking the most painfully sensitive area of the skin three times over 5 seconds at a rate of 1-2 cm/s with a Somedic brush. The patient will indicate the amount of pain evoked on a 100-millimeter visual analogue scale (VAS) by marking on a 100 mm line with the words "no pain" and "worst pain possible" on the left and right of it respectively. The position of the mark on the line from the left end to the right will be measured in millimetres to obtain level of dynamic mechanical allodynia (The higher the VAS score the more severe the dynamic mechanical allodynia). The change in dynamic mechanical allodynia will be assessed by comparing the scores obtained on trial day 1 versus day 14 and scores obtained on day 21 versus day 35.

SECONDARY OUTCOMES:
Analysis of pain relief | Scores will be obtained on trial day 14 and day 35.
  Pain relief measured on a 6-point categorical pain relief scale (0-worse pain to 5-complete pain relief). The higher the score the greater the pain relief.
Change in area of Punctate Hyperalgesia | Measurements will be performed on trial day 1, day 14 , day 21 and day 35.
  Area of punctate hyperalgesia will be obtained by marking and calculating the area of sensitivity to punctate stimulation of the skin with a Neuropen. Change in area of punctate hyperalgesia will be obtained by comparing the areas measured on trial day 1 versus trial day 14 and trial day 21 versus trial day 35.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ragavendran JV, Laferriere A, Xiao WH, Bennett GJ, Padi SS, Zhang J, Coderre TJ. Topical combinations aimed at treating microvascular dysfunction reduce allodynia in rat models of CRPS-I and neuropathic pain. J Pain. 2013 Jan;14(1):66-78. doi: 10.1016/j.jpain.2012.10.004. PMID 23273834
- [Background] Ragavendran JV, Laferriere A, Bennett GJ, Ware MA, Gandhi W, Bley K, Schweinhardt P, Coderre TJ. Effects of topical combinations of clonidine and pentoxifylline on capsaicin-induced allodynia and postcapsaicin tourniquet-induced pain in healthy volunteers: a double-blind, randomized, controlled study. Pain. 2016 Oct;157(10):2366-2374. doi: 10.1097/j.pain.0000000000000659. PMID 27385502
- [Background] Brown MB, Martin GP, Jones SA, Akomeah FK. Dermal and transdermal drug delivery systems: current and future prospects. Drug Deliv. 2006 May-Jun;13(3):175-87. doi: 10.1080/10717540500455975. PMID 16556569
- [Background] Li C, Sekiyama H, Hayashida M, Takeda K, Sumida T, Sawamura S, Yamada Y, Arita H, Hanaoka K. Effects of topical application of clonidine cream on pain behaviors and spinal Fos protein expression in rat models of neuropathic pain, postoperative pain, and inflammatory pain. Anesthesiology. 2007 Sep;107(3):486-94. doi: 10.1097/01.anes.0000278874.78715.1d. PMID 17721252
- [Background] Palos GR, Mendoza TR, Cantor SB, Aday LA, Cleeland CS. Perceptions of analgesic use and side effects: what the public values in pain management. J Pain Symptom Manage. 2004 Nov;28(5):460-73. doi: 10.1016/j.jpainsymman.2004.02.016. PMID 15504623
- [Derived] Fulas OA, Laferriere A, Ware DMA, Shir Y, Coderre TJ. The effect of a topical combination of clonidine and pentoxifylline on post-traumatic neuropathic pain patients: study protocol for a randomized, double-blind placebo-controlled trial. Trials. 2021 Feb 17;22(1):149. doi: 10.1186/s13063-021-05088-w. PMID 33596969